CLINICAL TRIAL: NCT06663475
Title: The Effectiveness of a Transtheoretical Model Based Health Education Intervention in Smoking Cessation Among Expectant Fathers: a Randomized Control Trial
Brief Title: A TTM-based Smoking Cessation Intervention in Helping Expectant Fathers to Quit Smoking and Maintain Abstinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Principle Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: L2023SYSU-HL-027; 72104259 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Smoking Cessation; Behavioral Intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- general health education videos (Active Comparator): general health education videos about hazards of secondhand smoke exposure for expectant fathers in obstetric clinic
  Interventions: Behavioral: usual care treatment
- TTM-based health education about smoking cessation tailored for expectant fathers (Experimental): health education videos based on transtheoretical model (TTM) to motivate quit attempt and maintain abstinence among smoking expectant fathers
  Interventions: Behavioral: TTM-based health education videos about smoking cessation for expectant fathers

INTERVENTIONS:
Behavioral: TTM-based health education videos about smoking cessation for expectant fathers — Tailored for expectant fathers, this smoking cessation health education information will be developed based on transtheoretical model to motivate a quit attempt and maintain abstinence by using videos.
  Arms: TTM-based health education about smoking cessation tailored for expectant fathers
Behavioral: usual care treatment — general health education videos about hazards of smoking for expectant fathers in obstetric clinic
  Arms: general health education videos

SUMMARY:
This study aims to evaluate the effectiveness of the video-based health education in smoking cessation among expectant fathers by using two-arm randomized clinical trial to motivate this subgroup attempt to quit, quit smoking and maintain abstinence in the long term.

ELIGIBILITY:
Inclusion Criteria:

* male adult
* has a pregnant partner
* at least smoke 1 cigarette per day on average in the last month
* be able to read or communicate in Chinese

Exclusion Criteria:

* be or was participated in other smoking cessation program in the past year
* mentally or physically unable to communicate with
* can't play videos by electronic devices
* the pregnant partner is a smoker

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1346 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence | 12 month follow-up after randomization
  Self-reported smoking abstinence will be biochemically validated by an exhaled carbon monoxide level < 4 parts per million (p.p.m) and negative for salivary cotinine test.

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 6, 12-month follow-up
  Subjects report that they had not smoked within the recent 7 days.
Smoking Reduction | end of intervention; 3,6,12 month after randomization
  Reduction in daily cigarette consumption by at least 50% compared with baseline.
Quit Attempt | end of intervention; 3,6,12 month after randomization
  Self-reported abstinence for at least 24 hours
The change in transtheoretical model stages | end of intervention; 3,6,12 month after randomization
  There are five stages according to the transtheoretical model, which are pre-contemplation (attempt to quit more than 30 days later), contemplation (attempt to quit within 30 days but more than 7 days), preparation (attempt to quit within 7 days), action stage (quitting) and maintain stage (maintain abstinence more than 6 months).
the Fagerstrom tolerance questionnaire | end of intervention; 3,6,12 month after randomization
  Nicotine Dependence will be measured by the Fagerstrom tolerance questionnaire.
Use of smoking cessation services | end of intervention; 3,6,12 month after randomization
  Smoking cessation services include nicotine replacement treatment, counseling for smoking cessation, telephone counselling and other services.
Biochemically validated smoking abstinence | 6 month follow-up
  self-reported smoking abstinence will be biochemically validated by an exhaled carbon monoxide level < 4 parts per million (p.p.m) and negative for salivary cotinine test.

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared one year after the results of the study'are published. The researchers can access the data by contacting the PI at xiaw23@mail.sysu.edu.cn with the research purpose described.
Supporting Information: SAP, Analytic Code
Time Frame: One year after the results of the study are published
Access Criteria: The researchers can access the data by contacting the PI at xiaw23@mail.sysu.edu.cn with the research purpose described.